CLINICAL TRIAL: NCT00476294
Title: Long-Term Observational Follow-Up Study of a Multicenter, Randomized, Double-Blind, Placebo-Controlled, Comparative Trial of AMD3100 (240 MCG/KG) Plus G-CSF (10 MCG/KG) Versus G-CSF (10 MCG/KG) Plus Placebo to Mobilize and Collect >/= 6 x 10^6 CD34+ Cells/KG in Multiple Myeloma Patients for Autologous Transplantation
Brief Title: Long-Term Follow Up Study for AMD3100 Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AnorMED (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-0665
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Disease-Free Survival; AMD3100; G-CSF; Autologous Transplantation
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: G + Placebo: G-CSF plus Placebo Arm (G + Placebo)
  Interventions: Other: Telephone Questionnaire
- Group 2: G + AMD3100: G-CSF plus AMD3100 Arm (G + AMD3100)
  Interventions: Other: Telephone Questionnaire

INTERVENTIONS:
Other: Telephone Questionnaire — Follow-Up Telephone Calls Every 6 Months for 5 Years.
  Other Names: Survey

SUMMARY:
Objectives:

The objective of this long-term observational study is to assess progression-free survival and overall survival for a period of five years following the first dose of study treatment (placebo or plerixafor [AMD3100]) in protocol AMD3100-3102. Patients that received at least 1 dose of study treatment (placebo or plerixafor) in the multicenter, randomized, double-blind, placebo-controlled AMD3100-3102 study, which was designed to evaluate plerixafor plus granulocyte colony stimulating factor (G-CSF) versus placebo plus G-CSF to mobilize hematopoietic stem cells for autologous transplantation of Multiple Myeloma (MM) patients are eligible.

DETAILED DESCRIPTION:
Informed Consent Process:

Your study doctor or staff will either meet with you in person or contact you by phone to review the study information. You will be given a copy of this consent form to review and ask questions.

If you agree to take part in this study, you should sign this consent form on the date that you agree to be in the study. If you agree to take part during a phone call with a member of the study team, you should sign and date the form right away, on the date of the phone call, and mail the form to the study doctor or staff. Please keep a copy for your own reference.

5-Year Follow-Up: You will be contacted by phone or in person at a visit, every 6 months for 5 years from the time of your first study drug/placebo dose in the 2004-0982 study. A placebo is a substance that looks like the study drug but has no active ingredients.

If you received a transplant in the 2004-0982 study, your first contact in this study will either be about 18 months from the time you began the 2004-0982 study, or at the time you sign this consent form.

If you did not receive a transplant, your first contact in this study will be at the time you sign this consent form.

At your first visit or call, you will be asked about the status of the disease, any changes in the multiple myeloma that may have occurred since the 2004-0982 study, and any additional treatments you may have received during that time.

At every visit or call after that, you will be asked about the status of the multiple myeloma, any changes in the disease, and any treatments you have received since the last visit or call. These questionnaires will take about 10 minutes each time.

Your doctor or the study staff also may contact your local doctor in order to collect information from your medical records or for information about your medical history and disease status.

Length of Study Participation:

You will be off study after your last study phone call or visit (about 5 years after your first study drug/placebo dose in the 2004-0982 study).

This is an investigational study. Up to 300 patients will participate in this multi-center study. Up to 12 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

* 1) All patients who received the study drug (placebo or plerixafor) on protocol AMD3100-3102 (2004-0982)

Exclusion Criteria: None

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were randomized in a double-blind study and received a stem cell transplant after treatment with AMD3100 and G-CSF OR treatment with Placebo and G-CSF.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival at 5 Years | 5 Years
  Progression-free survival defined as number of participants without disease progression at five years following the first dose of study treatment (placebo or plerixafor [AMD3100]).
Overall survival at 5 Years | 5 years
  Overall survival defined as number of participants alive after a period of five years following the first dose of study treatment (placebo or plerixafor [AMD3100]).

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org